CLINICAL TRIAL: NCT05682066
Title: TVMR With the Innovalve System Trial - Pilot in Georgia
Acronym: TWIST-PILOT-GE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INVL21-01-GE
Record Dates: First submitted 2022-12-22; First posted 2023-01-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Mitral Valve Regurgitation (Degenerative or Functional)
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Innovalve TMVR System (Experimental): MV replacement with Innovalve MR system
  Interventions: Device: Innovalve MR system

INTERVENTIONS:
Device: Innovalve MR system — Innovalve MR system

SUMMARY:
Study to evaluate the safety and performance of the Innovalve mitral valve replacement system

DETAILED DESCRIPTION:
The study is a multi-center, First-In-Human, prospective, single pilot study to evaluate the safety and performance of the Innovalve mitral valve replacement system

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant, symptomatic mitral regurgitation
* High risk for open-heart surgery
* Meets anatomical criteria

Exclusion Criteria:

* Unsuitable anatomy
* Patient is inoperable
* EF<25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Absence of implant or delivery related serious adverse events at 30 days | 30 days
  Absence of implant or delivery related serious adverse events

SECONDARY OUTCOMES:
Technical success | Procedure
  i. Absence of procedural mortality; and ii. Successful access, delivery, and retrieval of the device delivery system; and iii. Successful deployment and correct positioning of the first intended device; and iv. Freedom from emergency surgery or reintervention related to the device or access procedure.
Procedural success | 30 days
  All of the following must be present:
  I. Deployment of the device
  II. Absence of major device or procedure related serious adverse events, including:
  1. Death
  2. Stroke
  3. Life-threatening bleeding (MVARC scale)
  4. Major vascular complications
  5. Major cardiac structural complications
  6. Stage 2 or 3 acute kidney injury (includes new dialysis)
  7. Myocardial infarction or coronary ischemia requiring PCI or CABG
  8. Severe hypotension, heart failure, or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for 48 h.
  9. Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention
NYHA functional class | 30 days, 6, 1 year
Six-minute walk test | 30 days, 6, 1 year
Quality of life improvement (KCCQ-12) Kansas City Cardiomyopathy Questionnaire | 30 days, 6, 1 year
Reduction in Mitral Regurgitation grade | 30 days, 6, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No